CLINICAL TRIAL: NCT00796965
Title: A Phase I, Single-center, Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD7268 After Single Ascending Oral Doses in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of AZD7268 After Single Ascending Oral Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, M.D, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: D1151C00001
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Volunteer
Keywords: Phase 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD7268
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7268 — Solution/Capsule, Oral, once daily
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Single Ascending Dose Study

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Healthy male subjects and female subjects (of non-child bearing potential) with suitable veins for cannulation or repeated venipuncture

Exclusion Criteria:

* Inability to understand or cooperate with given information
* Positive human immune deficiency virus (HIV), Hepatitis B, or Hepatitis C test
* Clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology, and urinanalysis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-12; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single ascending dose administration of AZD7268 when given orally to healthy male subjects and female subjects of non-childbearing potential. | Safety assessments are made at each visit, at least daily, during the study.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD7268 in plasma and urine. | Blood and urine samples will be taken during the study.
To assess the effect of food on the safety and pharmacokinetic profile of AZD7268. | Safety assessments and blood and urine samples will be taken throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvan Hurewitz, M.D., Principal Investigator — AstraZeneca Clinical Pharmacology Unit, US
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States